CLINICAL TRIAL: NCT03206515
Title: The 18F Peel-way Sheath Versus the 18F Access Sheath With a Suction-evacuation Function MPCNL for the Management of 2-5cm Size Kidney Stones: A Randomized Controlled Trial
Brief Title: The 18F Peel-way Sheath Versus the 18F Access Sheath With a Suction-evacuation Function MPCNL for the Management of 2-5cm Size Kidney Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice President of the Hospital, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MRER(17)2016
Record Dates: First submitted 2016-10-27; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Renal Calculi
Keywords: Renal Pelvic Pressure
MeSH Terms: conditions — Kidney Calculi

ARMS (2):
- Group 1 (Other): Patients in Group 1 undergo Mini Percutaneous Nephrolithotomy with The 18F peel-way sheath group
  Interventions: Device: 18F Peel-Way Sheath
- Group 2 (Other): Patients in Group 2 undergo Mini Percutaneous Nephrolithotomy with The 18F access sheath with a suction-evacuation function group
  Interventions: Device: 18F access sheath with a suction-evacuation function

INTERVENTIONS:
Device: 18F Peel-Way Sheath — Patients undergoing Mini Percutaneous Nephrolithotomy with The 18F peel-way sheath
  Arms: Group 1
Device: 18F access sheath with a suction-evacuation function — Patients undergoing Mini Percutaneous Nephrolithotomy with The 18F access sheath with a suction-evacuation function
  Arms: Group 2

SUMMARY:
Percutaneous nephrolithotomy (PNL) has been considered as the first-line choice for the management of >20mm kidney stones. Microchannel percutaneous nephrolithotomy (Mini PCNL) which takes nephrolithotomy channel size less than or equal to 18, was first used in the treatment of children with kidney stones in 1997, then gradually applied to adult, aims to achieve the similar stone clearance rate as the standard channels, at the same time, reduce the complications. At present, the use of percutaneous renal surgery in our country is more than 18F plastic peel-away sheath, with the access sheath with a suction-evacuation function was first used by Guohua Zeng and so on. But there is still a lack of high quality evidence of Evidence-based medical evidence to compare the two kinds of sheath for the safety and effectiveness. Therefore, this study provides a reliable theoretical basis for the choice of the sheath for the treatment of 2-5cm size Kidney, and ultimately benefit patients with 20mm.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PNL) has been considered as the first-line choice for the management of >20mm kidney stones. Microchannel percutaneous nephrolithotomy (Mini PCNL) which takes nephrolithotomy channel size less than or equal to 18, was first used in the treatment of children with kidney stones in 1997, then gradually applied to adult, aims to achieve the similar stone clearance rate as the standard channels, at the same time, reduce the complications. At present, the use of percutaneous renal surgery in our country is more than 18F plastic peel-away sheath, with the access sheath with a suction-evacuation function was first used by Guohua Zeng and so on. But there is still a lack of high quality evidence of Evidence-based medical evidence to compare the two kinds of sheath for the safety and effectiveness. Therefore, this study provides a reliable theoretical basis for the choice of the sheath for the treatment of 2-5cm size Kidney, and ultimately benefit patients with 20mm.

ELIGIBILITY:
Inclusion Criteria:

* Patients consent for percutaneous renal stone removal
* Age 18 to 70 years
* Normal renal function
* ASA score Ⅰ and Ⅱ
* Renal stones 20-50mm

Exclusion Criteria:

* Patients with solitary kidney
* Uncorrected coagulopathy and active urinary tract infection (UTI)
* Morbid obese patients
* Patients who underwent transplant or urinary diversion
* Congenital abnormalities
* Patients will be excluded from the study if the undergoing standard PNL/mini-perc have purulent fluid in the initial puncture

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The renal pelvic pressure | During the procedure
  To measure the renal pelvic pressure during mini-PCNL procedure

SECONDARY OUTCOMES:
Perioperative complications | Intraoperatively or ≤ 1 month postoperatively
  Invaluate perioperative complications by modified Clavien system

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- epartment of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China